CLINICAL TRIAL: NCT00959985
Title: Early Detection and Intervention for Mild and Moderate Lymphedema in Patients Treated for Breast Cancer: A Randomized Trial
Brief Title: Early Detection and Intervention for Mild and Moderate Lymphedema in Patients Treated for Breast Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Chief of Breast Service, Radiation Oncology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-308; R01CA139118 (NIH)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema; Breast Cancer
Keywords: compression sleeve; compression bandage
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1A (No Intervention): Mild Lymphedema: Only required to meet with the lymphedema physical therapist
- Group 1B (Active Comparator): Mild Lymphedema: Fitted for compression sleeve
  Interventions: Device: Compression Sleeve
- Group 2A (Active Comparator): Moderate lymphedema: Fitted with a compression sleeve
  Interventions: Device: Compression Sleeve
- Group 2B (Active Comparator): Moderate Lymphedema: Fitted with compression sleeve and instructed to wear a short-stretch compression bandage
  Interventions: Device: Compression Sleeve; Device: Short-Stretch Compression Bandage

INTERVENTIONS:
Device: Compression Sleeve — Worn for a minimum of 12 hours per day
  Arms: Group 1B; Group 2A; Group 2B
Device: Short-Stretch Compression Bandage — Worn overnight at least 5 nights of the week
  Arms: Group 2B

SUMMARY:
Women who have been treated for breast cancer may be at risk for lymphedema or arm swelling. Currently, there are no clear treatment guidelines for lymphedema. One treatment method used to treat lymphedema is the use of compression sleeves to encourage the flow of lymph fluid out of the arms and prevent arm swelling in the future. Another treatment method is more intensive and involves wearing compression sleeves as well as special compression bandages overnight. It is unclear whether the use of compression with both sleeves and bandaging is more effective in treating lymphedema than the use of compression sleeves alone. The purpose of this research study is to evaluate the effectiveness of the use of compression garments in preventing or slowing the progression of lymphedema in breast cancer patients.

DETAILED DESCRIPTION:
* Because no one knows which of the study options is best, participant's will be randomized into one of the study groups. Participants with mild lymphedema will be randomized into either Group 1A or Group 1B. Participants with moderate lymphedema will be randomized into either Group 2A or Group 2B.
* All study participants will meet with a lymphedema physical therapist to review daily shoulder range of motion exercises to help minimize their arm swelling. They will be asked to record their range of motion exercises and activities in a study treatment journal. Participants will bring their journal to each study visit (every 4 weeks).
* Group 1A will only be required to meet with the lymphedema physical therapist as described above.
* Group 1B and Group 2A will be fitted with a compression sleeve at their first lymphedema physical therapy visit. They will wear the sleeve for a minimum of 12 hours per day.
* Group 2B will also be fitted with a compression sleeve at their first lymphedema physical therapy visit and will wear the sleeve for a minimum of 12 hours per day. They will also be instructed to wear a short-stretch compression bandage that goes from the top of the hand to the armpit. They will be asked to wear this compression bandage during the night. The overnight compression bandage should be worn for at least 5 nights out of the week.
* Participants will come to the clinic every 4 weeks. The following tests and procedures will be performed: height and weight measurements; review of any side effects; arm volume measurements for both arms; questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive or in-situ carcinoma of the breast
* Participants must have undergone sentinel lymph node mapping or axillary dissection
* Participants must have had a pre-operative Perometer measurement, and consecutive measurement at 4-6 month intervals prior to the onset of low volume edema (>5% from baseline)
* Age > 18 years
* Life expectancy of greater than 1 year
* Participants must have a Perometer measurement of 5% or greater volume difference (RVC) to qualify for randomization
* Ability to understand and willingness to sign a written informed consent document
* Willingness to comply with required follow up Perometer measurements and clinical visits

Exclusion Criteria:

* Known metastatic disease or other locally advanced disease in the thoracic or cervical regions
* Any patient who will not be returning routinely for follow-up
* Known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of primary lymphedema
* History of prior surgery or radiation to the head, neck, upper limb, or trunk
* Evidence that axillary lymph node malignancy is causing lymphedema due to recurrence as per physician discretion
* Any patient who has bilateral lymph node mapping or dissection
* Any patient with a current case of cellulitis
* Patients with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancer are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G. Taghian, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Started | 8 | 7 | 4 | 4
Completed | 8 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B | Total
Number analyzed (Participants) | 8 | 7 | 4 | 4 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 3 | 17
  >=65 years | 3 | 2 | 0 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 4 | 4 | 23
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Identify the Number of Patients Who Experienced Reduction in Edema With Compression Garment Usage for Low Volume Lymphedema Associated With Breast Cancer Treatment
Description: Participants who are randomized to receive compression treatment will have their arm volume measured at regular intervals throughout the study period. Participants' arm volume, as measured by the validated Relative Volume Change (RVC) equation, at the end of the intervention period will be assessed to determine the efficacy of the compression garment intervention and whether or not it was successful in reducing the participants' arm edema to RVC<10%.Data was collected in study participants enrolled in Group 1A and Group 1B only (15 patients total), and the percentage of participants who experienced reduction in edema is reported below.
Time Frame: 5 years
Population: This outcome measure was compared between Group 1A (control) and Group 1B (compression garment). No data was collected for this outcome in Groups 2A and 2B
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 8 | 7 | 0 | 0
Participants | 7 | 4 |  |

2. Primary Outcome: To Identify the Number of Patients Who Experienced Reduction in Edema With Compression Garments +/- Night Compression Bandaging for Moderate Volume Lymphedema Due to Breast Cancer Treatment
Description: Participants who are randomized to receive compression treatment with/without night bandaging will have their arm volume measured at regular intervals throughout the study period. Participants' arm volume, as measured by the validated Relative Volume Change (RVC) equation, at the end of the intervention period will be assessed to determine the efficacy of the compression garment intervention and whether or not it was successful in reducing the participants' arm edema to RVC<10%. Data was collected in participants enrolled in Group 2A and 2B only (8 participants total), and the percentage of participants who experienced reduction in edema is reported below.
Time Frame: 5 years
Population: This outcome measure was compared between Groups 2A and 2B. No data was collected for Group 1A and 1B as this outcome does not apply to these groups
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 0 | 0 | 4 | 4
Participants | 0 | 0 | 2 | 3

3. Primary Outcome: To Assess Survey Response Scores Regarding Symptoms Associated With Varying Degrees of Lymphedema
Description: Symptoms were assessed through the Lymphedema Evaluation Following Treatment of Breast Cancer (LEFT-BC) survey. The responses were scored on a scale from 0-51, where higher score was associated with presence of more symptoms (0=no symptoms, 51 = most symptoms)
Time Frame: 5 years
Population: Median scores of the symptom-related questions on the LEFT-BC survey, per group, are indicated below. Participants who did not complete or return surveys due to non-compliance were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 5 | 7 | 2 | 1
units on a scale | 4 [3.25 to 10] | 6.46 [1 to 20] | 6.58 [5.5 to 7.67] | 2.4 [2.4 to 2.4]

4. Primary Outcome: To Assess Survey Response Scores Regarding Fear Avoidance Behavior Associated With Varying Degrees of Lymphedema
Description: Fear avoidance behavior was assessed through the Lymphedema Evaluation Following Treatment of Breast Cancer (LEFT-BC) survey. Participant responses were scored on a scale from 7-28, where higher score was associated with higher level of fear of using arm (7= least fear level; 28= most fear level)
Time Frame: 5 years
Population: Median scores for the fear avoidance behavior section on the LEFT-BC survey, per group, are indicated below. Participants who did not complete or return surveys due to non-compliance were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 5 | 7 | 2 | 1
units on a scale | 13.3 [10 to 20.25] | 16.5 [12.67 to 19.4] | 20.75 [19.67 to 21.8] | 17 [17 to 17]

5. Primary Outcome: To Assess Survey Response Scores Regarding Quality of Life as it Associated With Varying Degrees of Lymphedema
Description: Quality of life was assessed through the Lymphedema Evaluation Following Treatment of Breast Cancer (LEFT-BC) survey. Participant responses were scored on a scale from 0-141, where higher score was associated with higher post-operative quality of life (0= worst; 141= best)
Time Frame: 5 years
Population: Median scores for the quality of life questions on the LEFT-BC survey, per group, are indicated below. Participants who did not complete or return surveys due to non-compliance were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 5 | 7 | 2 | 1
units on a scale | 102.5 [89.25 to 124.8] | 110 [98.1 to 128] | 99.17 [90.5 to 107.8] | 106.8 [106.8 to 106.8]

6. Primary Outcome: To Assess Survey Response Scores Regarding Upper Extremity Function as it Associated With Varying Degrees of Lymphedema
Description: Upper extremity functions were assessed through the Lymphedema Evaluation Following Treatment of Breast Cancer (LEFT-BC) survey. Participant responses were scored on a scale from 19-95, where higher score was associated with more difficulty utilizing arm for daily activities (19 = least difficulty; 95 = most difficulty)
Time Frame: 5 years
Population: Median scores for the upper extremity function questions on the LEFT-BC survey, per group, are indicated below. Participants who did not complete or return surveys due to non-compliance were excluded from this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 5 | 7 | 2 | 1
units on a scale | 21.2 [14.25 to 49.25] | 24.5 [19 to 43.5] | 24.8 [22.8 to 26.8] | 19.6 [19.6 to 19.6]

7. Secondary Outcome: To Identify the Number of Patients With Risk Factors Associated With the Onset of Lymphedema That Are Both Related and Unrelated to Treatment for Breast Cancer
Description: Surgical and radiation therapy risk factors for lymphedema (surgery to lymph nodes, radiation to lymph nodes), as well as risk factors unrelated to breast cancer treatment such as high BMI were collected upon medical record review
Time Frame: 5 years
Population: The number and percentage of participants in each group who had at least 2 known risk factors for lymphedema is documented in the outcome measure data table below
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 8 | 7 | 4 | 4
Participants | 4 | 6 | 2 | 4

8. Secondary Outcome: To Evaluate the Number of Patients With Low-level Arm Swelling in Order to Understand the Natural History of Lymphedema After Treatment for Breast Cancer
Description: We recorded the number of participants who had low-level arm swelling, as defined by the Relative Volume Change (RVC) equation of >5%-<10%, at the time of their post-operative follow up to determine if women who had low-level arm swelling were more likely to develop lymphedema
Time Frame: 5 years
Population: Number and percentage of participants who had low-level arm swelling at their post-operative follow up are documented below
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
Number analyzed (Participants) | 8 | 7 | 4 | 4
Participants | 3 | 2 | 2 | 2

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group 1A | Group 1B | Group 2A | Group 2B
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/8 | 3/7 | 2/4 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1A (N=8) | Group 1B (N=7) | Group 2A (N=4) | Group 2B (N=4)
Arm lymphedema progressed beyond allowed study parameters (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) — Participants who experienced an increase in arm volume >10% and did not wish to be re-randomized were removed from study and treated at discretion of physical therapist. They remained on active lymphedema screening at treating institution
Periodic mild pain while wearing compression garments (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One participant experienced periodic mild pain while wearing compression garments. The physical therapist advised the participant to not wear the garments when they were causing her pain; participant continued study without further complication
Presence of symptoms (e.g. swelling, tightness) in arm after completion of treatment period (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — After completing study requirements 1 participant contacted the physical therapist (PT) to report feeling more symptoms in the arm. The PT determined her symptoms were related to her cording, not lymphedema, and recommended stretching exercises.
Symptoms of leg edema prior to study enrollment date (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — One participant experienced increased leg swelling and then underwent a lower-extremity venous ultrasound to rule out blood clot.This was negative and the protocol treatment she received for breast cancer-related lymphedema was not interrupted

LIMITATIONS AND CAVEATS:
This trial was terminated due to slow accrual and small number of subjects for whom data was collected (23 out of expected 334). Study did not reach statistical power to conduct detailed analysis, results should be interpreted with this in mind

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes